CLINICAL TRIAL: NCT03979105
Title: Cardiovascular and Neuropsychiatric Side Effects in Ketamine Analgesic Infusions in Acute Pain
Brief Title: Cardiovascular Safety After Continuous Ketamine Infusion
Status: Completed | Type: Observational
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Other Study IDs: UdeA1005
Record Dates: First submitted 2019-04-04; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Pain; Ketamine Adverse Reaction; Postoperative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ketamine infusion: Ketamine infusion treatment for acute pain in adult population in all type of surgery that received adjuvant analgesia with ketamine 0.1mg/kg/h during 48 hours.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Drug: Ketamine Side effects associated with ketamine infusion to treat acute pain, were reviewed after 48 hours of exposure and frequency of tachycardia, hypertension, hallucinations, delirium and nightmares were registrated for comparison
  Other Names: Ketalar

SUMMARY:
Observational study that evaluate the cardiovascular and neuropsychiatric side effects of ketamine analgesic infusions for acute pain

DETAILED DESCRIPTION:
Severe acute pain and opioid tolerance is an important symptom in patients after surgery.

Ketamine in analgesic infusion has been described to decrease acute pain, in patients with opioid tolerance. Ketamine use has been associated with side effects, which are doses dependant. Those side effects are mainly cardiovascular: Hypertension, tachycardia, and neuropsychiatric: delirium, hallucinations,nightmares that potentially compromise recovery of patients.

Objective:

To determine retrospectively in data bases the frequency of tachycardia, hypertension, delirium, hallucinations and nightmares, in adult patients that received ketamine infusions before and after administration of this drug in the first 48 hours to treat acute and postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Acute and Postoperative pain
* Ketamine infusion at 0.15 mg/kg/h or below

Exclusion Criteria:

* Cognitive disfunction psychiatric illness
* Acute cardiovascular disease
* Anemia with Hb less than 7 g/dl
* Decompensated hyperthyroidism
* Low cardiac output
* Incomplete medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with acute pain after surgery or medical painful condition
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Tachycardia | 2 days
  Presence of absence of tachycardia (100 or above beats for minute) as physiological parameter recorded with cardioscope in the first 48 hours in clinical chart database after the infusion of ketamine has started.
Hypertension | 2 days
  Presence or absence of hypertension (140/90 mm Hg or above ) as physiological parameter recorded with electronic arm manometer in the first 48 hours in clinical chart database after the infusion of ketamine has started.

SECONDARY OUTCOMES:
Delirium | 2 days
  Presence of absence of delirium reported in clinical records electronic database by nurse or physician in the first 48 hours after the infusion of ketamine has started.
Hallucinations | 2 days
  Presence of absence hallucinations reported in clinical electronic database records by nurse or physician in the first 48 hours after the infusion of ketamine has started.
Nightmares | 2 days
  Presence of absence of nightmares reported in clinical electronic database records by nurse or physician, in the first 48 hours after the infusion of ketamine has started.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Cadavid, MD, Principal Investigator — Anesthesiology Investigator
Locations (2):
- Colombia (2):
  - hospital universitario San Vicente Fundacion, Medellín, Antioquia
  - Adriana Cadavid, MD, Medellín, Antiquia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avidan MS, Fritz BA, Maybrier HR, Muench MR, Escallier KE, Chen Y, Ben Abdallah A, Veselis RA, Hudetz JA, Pagel PS, Noh G, Pryor K, Kaiser H, Arya VK, Pong R, Jacobsohn E, Grocott HP, Choi S, Downey RJ, Inouye SK, Mashour GA. The Prevention of Delirium and Complications Associated with Surgical Treatments (PODCAST) study: protocol for an international multicentre randomised controlled trial. BMJ Open. 2014 Sep 17;4(9):e005651. doi: 10.1136/bmjopen-2014-005651. PMID 25231491
- [Background] Kase D, Imoto K. The Role of HCN Channels on Membrane Excitability in the Nervous System. J Signal Transduct. 2012;2012:619747. doi: 10.1155/2012/619747. Epub 2012 Aug 13. PMID 22934165
- [Background] Pomeroy JL, Marmura MJ, Nahas SJ, Viscusi ER. Ketamine Infusions for Treatment Refractory Headache. Headache. 2017 Feb;57(2):276-282. doi: 10.1111/head.13013. Epub 2016 Dec 27. PMID 28025837
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642
- [Background] Radvansky BM, Shah K, Parikh A, Sifonios AN, Le V, Eloy JD. Role of ketamine in acute postoperative pain management: a narrative review. Biomed Res Int. 2015;2015:749837. doi: 10.1155/2015/749837. Epub 2015 Oct 1. PMID 26495312
- [Background] Garg N, Panda NB, Gandhi KA, Bhagat H, Batra YK, Grover VK, Chhabra R. Comparison of Small Dose Ketamine and Dexmedetomidine Infusion for Postoperative Analgesia in Spine Surgery--A Prospective Randomized Double-blind Placebo Controlled Study. J Neurosurg Anesthesiol. 2016 Jan;28(1):27-31. doi: 10.1097/ANA.0000000000000193. PMID 26018671
- [Background] Assouline B, Tramer MR, Kreienbuhl L, Elia N. Benefit and harm of adding ketamine to an opioid in a patient-controlled analgesia device for the control of postoperative pain: systematic review and meta-analyses of randomized controlled trials with trial sequential analyses. Pain. 2016 Dec;157(12):2854-2864. doi: 10.1097/j.pain.0000000000000705. PMID 27780181
- [Derived] Cadavid AM, Casas FD, Camelo JE, Tovar A, Ramirez CD, Calle E, Visbal K. Effect of Analgesic Low-Dose Ketamine Infusions on the Cardiovascular Response: A Retrospective Analysis. Pain Physician. 2023 Sep;26(5):495-502. PMID 37774188